CLINICAL TRIAL: NCT02214381
Title: A Prospective, Multicenter, Open-label Comparison of Pre-surgical Myocet/ Cyclophosphamide (MC) q3w Followed by Either MC or Paclitaxel - Depending on Early Response Assessment by Ultrasound or by Toxicity for Elderly Non Frail Primary Breast Cancer Patients With Increased Risk of Relapse.
Brief Title: A Prospective, Multicenter, Open-label 12 Week Neoadjuvant Phase II Trial Optimizing Taxane Therapy in Elderly Patients With Low Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM06 / ADAPT Elderly
Record Dates: First submitted 2014-07-31; First posted 2014-08-12 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Early Primary Breast Cancer
Keywords: breast cancer; elderly
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycet/Cyclophosphamid (Active Comparator): 4 x Myocet 60 mg/m² q3w in combination with 4 x cyclophosphamide 600 mg/m² q3w depending on early response assessment by ultrasound or on toxicity profile.
  Interventions: Drug: Myocet; Drug: Cyclophosphamide
- Myocet/Cyclophosphamide/Paclitaxel (Active Comparator): 2 x Myocet 60 mg/m² q3w in combination with 2 x cyclophosphamide 600 mg/m² q3w followed by 6 x paclitaxel 80 mg/m² q1w depending on early response assessment by ultrasound or on toxicity profile.
  Interventions: Drug: Myocet; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Myocet
  Other Names: Doxorubicin
Drug: Cyclophosphamide
Drug: Paclitaxel
  Arms: Myocet/Cyclophosphamide/Paclitaxel

SUMMARY:
Comparison of pre-surgical Myocet/ Cyclophosphamide (MC) q3w followed by either MC or Paclitaxel - depending on early response assessment by ultrasound or by toxicity for elderly non frail primary breast cancer patients with increased risk of relapse.

ELIGIBILITY:
General Inclusion Criteria for ADAPT:

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Candidate for chemotherapy on the basis of conventional criteria
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4a-c
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology)
* Tumor block available for central pathology review
* Performance Status ECOG <= 1 or KI >= 80%
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up
* Patients must qualify for neoadjuvant treatment
* LVEF > 50%; LVEF within normal limits of each institution measured by echocardiography and normal ECG (within 42 days prior to chemotherapy)

  * Laboratory requirements :

    * Leucocytes ≥ 3.5 x 109/L
    * Platelets ≥ 100 x 109/L
    * Hemoglobin ≥ 10 g/dL
    * Total bilirubin ≤ 1 x ULN
    * ASAT (SGOT) and ALAT (SGPT) ≤ 2.5 x UNL
    * Creatinine ≤ 175 µmol/L (2 mg/dl)

Additional inclusion criteria ADAPT Elderly:

* ≥ 70 years old
* Charlson scale ≤ 2
* HR+/HER2- disease: if RS and sequential testing are available N0-1/RS 12-25/poor response or N0-1/RS ≥26
* All G3 with Ki-67 ≥40% in tumors >1cm
* All N2
* All TN
* All subtypes

General Exclusion Criteria for ADAPT:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry (concurrent participation in non-interventional post authorization safety studies not influencing the primary study endpoints is allowed, e.g. WSG PROTROCA for evaluation of primary/secondary G-CSF prophylaxis)
* Male breast cancer
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Patient not able to consent

Additional Exclusion Criteria ADAPT Elderly:

* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study
* Inadequate organ function (e.g. hepatic impairment, pulmonary disease, etc.)
* Uncompensated cardiac function (current unstable ventricular arrhythmia requiring treatment, history of symptomatic CHF NYHA classes II-IV), history of myocardial infarction or unstable angina pectoris within 12 months of enrollment, history of severe hypertension, CAD - coronary artery disease)
* Severe dyspnea
* Pneumonitis
* Abnormal blood values:
* Thrombocytopenia > CTCAE grade 1
* Increases in ALT/AST > CTCAE grade 1
* Hypokalaemia > CTCAE grade 1
* Neutropenia > CTCAE grade 1
* Anaemia > CTCAE grade 1

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of pCR rates in patients with early response and no severe toxicity (Group 1) and in other patients (Group 2). | After 5 years of follow-up.

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) after 1 x MC in patients with primary prophylaxis (PP) vs. others. | After 5 years of follow-up.
Toxicity in the 4 x MC versus 2 x MC followed 6 x Pac arm as measured by adverse events. | After 5 years of follow-up.
Number of pCR in non-responders to MC. | After 5 years of follow-up.
G-CSF use in terms of primary or secondary prophylaxis per patient including occurence febrile neutropenia per patient per cycle | After 5 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (2):
- Germany (2):
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach
  - Breast Center of the University of Munich (LMU) Universitätsfrauenklinik Großhadern, Munich